CLINICAL TRIAL: NCT04115579
Title: The Impact of Low Glycaemic Index (GI) Biscuits on Postprandial Glycaemia Using the Continuous Glucose Monitoring System (CGMS™) (Biscuit Study (BIS) Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018/01066
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biscuit 1 Control (Experimental): Consumption of control biscuit for breakfast and afternoon snack and impact on postprandial glucose and insulin
  Interventions: Other: Biscuit 1 Control
- Biscuit 2 Test (Experimental): Consumption of test biscuit for breakfast and afternoon snack on postprandial glucose and insulin
  Interventions: Other: Biscuit 2 Test

INTERVENTIONS:
Other: Biscuit 1 Control — Consumption of control biscuit of a higher glycaemic index at one session during breakfast and afternoon snack
  Arms: Biscuit 1 Control
Other: Biscuit 2 Test — Consumption of test biscuit of a lower glycaemic index at one session during breakfast and afternoon snack
  Arms: Biscuit 2 Test

SUMMARY:
To investigate whether low glycaemic index (GI) biscuits have the greatest impact on the post-meal glucose response and on the overall 24 hour blood glucose control, using the continuous glucose monitoring system (CGMS™)

DETAILED DESCRIPTION:
The study was a randomized, non-blinded, crossover design. Randomization conducted using www.randomizer.org. Each participant came for two test sessions (each of 3 days- Days 0, 1 and 2) with each session separated by at least three days (to avoid crossover effects). Test foods: The foods were Control and Test [Low glycemic index (GI)] biscuits. The foods will vary in macronutrient, micronutrients and fibre contents. Screening session: Potential participants attend a first session for consenting and screening procedures. Subjects will be at the centre for the study between 8:00-9:00am, with screening session lasting approximately 1 hour. Subjects will have to come following a 10-12 hour overnight fast each day. Fingerprick blood sample (5μl) is required for the screening session (to establish fasting glucose concentration). Screening questionnaire: The screening questionnaire will include contact information, demographic, general health details, and physical activity level. This information will be used to determine whether the participant is eligible for the study, as well as to check for any possible confounders that may influence the study outcomes. Anthropometric measurements: Body weight and body composition will be measured using bioelectrical impedance analysis (Tanita scale). Height will be measured using a stadiometer in order to calculate participants' BMI. Waist circumference will be measured at the minimum circumference between the iliac crest and the rib cage. Hip circumference will be measured at the maximum protuberance of the buttocks. Biceps and triceps skinfold measurements will also be taken. Blood pressure will also be measured. Blood pressure: Blood pressure will be measured using an Omron blood pressure monitor (Model HEM-907) at baseline. Participants will be seated for five minutes before blood pressure is measured. Measurements will be taken in duplicate and the averaged results will be recorded. (approximately 1 teaspoon or 5 ml) will be collected from subject via passive drooling (only once during). Start of test session (Day 0-Day 2) Day 0 If subject is eligible, subjects will be enrolled into the study. Subject will undergo the insertion of the Continuous Glucose Monitoring System (CGMS™) sensor the day before the test day (Day 0) to allow for the monitor to stabilize overnight. Medtronic's iPro2 Professional CGMS, designed to gain more complete insights into the glycaemic profiles of a person. The CGMS sensor will be inserted into the adipose tissue in the abdominal area by trained researchers and nurses. Subjects will have to wait in the laboratory for 1 hour after insertion for the sensor to be stabilized. After 1 hour the inserted CGMS sensor will be calibrated against a manual finger-prick blood glucose sample (5 μL, a small drop). Manual calibration using finger-prick blood samples will need to be carried out before every meal and before bed in the night (5 μL each for before dinner and before sleeping). The calibrations before dinner and bed will have to be carried out the subjects at home. Therefore, the subjects will be provided with a finger-prick blood glucose test kit to take home and instructed on how to correctly use it and measure blood glucose values. Calibration finger pricks will be made using disposable individual lancets. This may cause minimal discomfort. The volume of blood taken each time will be 5 μL (a small drop). For Day 0, subjects will be provided a standard dinner meal to be consumed at home at 7pm. Afterwhich, they will be asked to not eat and drink anything except water after 10:30 pm. They will also be instructed to arrive at the CNRC the following morning in an overnight fasted state. On the evenings before the test sessions, subject will be reminded to have no strenuous physical activities and no consumption of alcoholic beverages. Day 1 On the test Day 1, participants will be asked to attend the testing sessions after an overnight fast of ten to twelve hours, and arrive between 8:00-9:00am, with each session lasting approximately 4 hours. One fasting blood sample will be collected by fingerprick for calibration of the CGMS glucose meter (5 μL, a small drop). Then, an indwelling catheter will be inserted into a vein in the forearm. Subsequently, a blood sample will be taken from a cannula to measure baseline values. Immediately after that, participants will be served a test breakfast, where they will be asked to consume within 15 minutes. Following the test breakfast meal, further blood samples will be taken (from the cannula) for the next 15, 30, 45, 60, 90, 120, 150, 180 minutes. The blood samples collected at each timepoint will be measured for insulin and metabolic biomarkers related to the intake of the test meal ingredients. The amount of blood that will be collected at every time point will be about 1.2 teaspoon of blood (approximately 6 ml), the accumulative amount per test session will not be more than 11 teaspoons of blood (approximately 55 ml), and the accumulative amount for the entire study duration will not be more than 22 teaspoons of blood (approximately 110 ml), by cannula. For the fingerprick calibration, 5 μL is taken after insertion of sensor, before each meal and before sleeping. So a total of 9 fingerpricks will be taken for one test session. Therefore, a total of 18 fingerpricks for the entire two sessions. (approximately 90 μL equivalent to approximately 1/5 of a teaspoon). A standard lunch will then be served and afterwhich the cannula is removed. Subjects will take a fingerprick blood glucose (5 μL, a small drop) for calibration of the CGMS before their standard lunch meal. Subjects are to consume the entire lunch meal in 15 minutes. After lunch, participants will be provided with their snack and dinner meal to be consumed at home and they will leave the research facility. Before snack, dinner and before sleeping, participants are to take their own fingerprick blood glucose for calibration of the CGMS.Day 2 Participants will return the following day, Day 2, between 8:00-9:00am. Participants will have the CGMS sensor removed. A final fingerprick (5 μL, a small drop) for calibration purposes will be done 15 minutes before removal of the sensor. This marks the end of one session and participant will return for the next session after 3 days of washout period. Participants attend a total of about 15 hours for two sessions (including one screening visit lasting around 1 hour). Participants will spend approximately 1 hour for screening session, 1 hour for Day 0, 4 hours for Day 1 and about half hour on Day 2. This will repeat for the next session. All test and standard meals in the research facility will be served with 250ml of water. All the study diets will be prepared in the CNRC food preparation kitchen and will use locally sourced ingredients and food purchased from local supermarkets and food distributors.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Healthy Asian Chinese
* Aged between 21 - 40 years
* Body mass index between 18.5 to 25.0 kg/m2
* Normal blood pressure <140/90 mmHg
* Fasting blood glucose <6.0 mmol/L

Exclusion Criteria:

* Smoking
* Allergic/intolerant to any of the test foods to be administered, or any of the following common food and ingredients: eggs, fish, milk, peanuts, and tree nuts, shellfish, soya, wheat, gluten, cereal, fruits, dairy products, meat, vegetable, sugar and sweetener, natural food colourings or flavourings, etc.
* Anyone with intentional food restrictions
* People with known glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* Having metabolic or cardiovascular diseases (such as diabetes, hypertension, heart condition, etc), Having any other diseases involving the small intestine or the colon (e.g., irritable bowel syndrome, inflammatory bowel disease, gastric reflux) or having any liver or kidney disorders or any family history of kidney stones
* Having medical conditions and/or taking medications known to affect glycemia (glucocorticoids, thyroid hormones, thiazide diuretics)
* Taking any prescribed medication or dietary supplements which may interfere with the study measurements
* Excessive alcohol consumption: consuming ≥ 6 alcoholic drinks per week
* Individuals who have donated blood or taken part in other studies within 4 weeks of study participation.
* Have poor veins impeding venous access
* Have history of severe vasovagal syncope (blackouts or near faints) following blood draws
* Have known Chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Have active Tuberculosis (TB) or currently receiving treatment for TB
* Individuals who partake in sports at the competitive and/or endurance levels.
* A team member of the study or is an immediate family member (Immediate family defined as a spouse, parent, child, or sibling, whether biological or legally adopted

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male volunteers
Enrollment: 14 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose | Up to 24 hours
  Glucose measurements taken using the Continuous Glucose Monitoring System

SECONDARY OUTCOMES:
Postprandial insulin | up to 180 minutes
  Plasma blood will be analyzed using COBAS

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No